CLINICAL TRIAL: NCT02529306
Title: The Correlation Between Testosterone and Cortisol Level and Inflammatory Markers Levels in Type 2 Diabetic Men.
Acronym: BZMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0045-15BNZ
Record Dates: First submitted 2015-07-29; First posted 2015-08-20 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetic
Keywords: men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- two parallel group: group with inflammatory markers high levels and control group with inflammatory normal levels markers.

SUMMARY:
Many type 2 diabetic men have low serum testosterone levels. Our aim in this trial is to check if there is a correlation between serum or hair testosteron levels and serum or hair cortisol levels in type 2 diabetic men. We'll also examine whether there is a correlation between serum and hair testosterone levels and cortisol levels and serum inflammatory markers.

If such correlation will be found- then it is possible that excess cortisol or an abnormal inflammatory status- may cause the low testosterone levels that seen in type 2 diabetic men.

DETAILED DESCRIPTION:
Eligible participants are type 2 diabetic men who visit our clinic, as part of their routine medical surveillance, and other 10 healthy volunteers (men) as a control group.

All the participants will sign an informed consent form. The study will include 30 type 2 diabetic men, (40-55 years old) and 10 healthily volunteers (same age group).

In addition to routine blood test of blood count, kidney function and liver enzymes will be taken blood samples of total testosterone serum levels, total cortisol serum levels and serum inflammation markers levels, and also a sample of head-hair for cortisol and testosterone levels (1 cm of occipital hair weighing 50 mg).

Optional: from patients who will agree to visit the clinic after 8 hours-fast will be also taken one additional blood sample of fasting glucose, insulin and C-peptide levels, in order to estimate their insulin resistance status, and it's possible correlation to the other measures.

From the 10 healthy volunteers In addition will be taken blood and hair samples of the above parameters, as a control.

ELIGIBILITY:
Inclusion Criteria:

* men age 40-55
* type 2 diabetic

Exclusion Criteria:

* HIV
* septic disease

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Type 2 diabetic men, age 40-55
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Testosterone level | 24 months
  single blood and hair sample will be drawn to measure Testosterone levels (nmol/L)
Cortisol level | 24 months
  single blood and hair sample will be drawn to measure cortisol levels (mcg/dl)
C-reactive protein levels | 24 months
  single blood sample will be drawn to measure c-reactive protein levels (mcg/dl)
Anti Tumor Necrosis Factor alpha | 24 months
  single blood sample will be drawn to measure Anti Tumor Necrosis Factor alpha levels (pg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Haifa, Israel